CLINICAL TRIAL: NCT02988999
Title: The Efficacy of D-allulose (Psicose) on Weight and Fat Loss and Insulin Resistance by a Randomized Double-blind, Parallel-group Study in Non-diabetic Obese Subjects
Brief Title: Efficacy of D-allulose on Weight and Fat Loss and Insulin Resistance in Non-diabetic Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Collaborators: Kagawa University (Other)
Responsible Party: Principal Investigator, Supawan Buranapin, Assisstant professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMU-D-allulose02
Record Dates: First submitted 2016-11-21; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: D-allulose or erythritol
MeSH Terms: conditions — Obesity | interventions — Erythritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-allulose (Experimental): D-allulose 5 gm 3 times a day
  Interventions: Dietary Supplement: D-allulose
- erythritol (Active Comparator): erythritol 5 gm 3 times a day
  Interventions: Dietary Supplement: erythritol

INTERVENTIONS:
Dietary Supplement: D-allulose — D-allulose (psicose), a C-3 epimer of D-fructose, is defined one of the rare sugars since it is rarely found in nature. Rare sugars are monosaccharides which present in small quantities in commercial mixtures of D-glucose and D-fructose obtained from hydrolysis of sucrose or isomerization of D-glucose (5). D-allulose (psicose) has been demonstrated to be a non-calorie monosaccharide which has approximately 70% sweetness of sucrose. Various physiological activities of D-allulose (psicose) have been revealed. Of those, its glucose suppressive effect has been proven by both animal and clinical studies.
  Arms: D-allulose
Dietary Supplement: erythritol — non-calorie sweetener
  Arms: erythritol

SUMMARY:
Prospective, randomized, double-blind, controlled-trial 30 subjects in each groups Group - I consume pure D-allulose 5 g 3 times a day before meal to right after meal (with any liquid) and Group - II control group with non-calorie sweetener erythritol 5 g 3 times a day before meal to right after meal (with any liquid) Total number: n = 60 Either males or females, non-diabetic, aged > 18 years old with BMI ≥ 25 kg/m2

Primary objectives Efficacy

1. Compare the efficacy of pure D-allulose (psicose) plus conventional therapy on 1.1 visceral fat area (VFA), subcutaneous fat area (SFA), total fat area (TFA) change 1.2 body weight, BMI and body fat percentage (with impedance method) change after 24 weeks of D-allulose (psicose) consumption to erythritol consumption and between pre- and post-intervention.

Secondary objectives 1. Efficacy of pure D-allulose (psicose) plus conventional therapy versus erythritol plus conventional therapy on 1.1 insulin resistance, fasting plasma glucose, HbA1c 1.2 adiponectin, leptin and tumor necrosis factor-alpha, lipid profiles (total cholesterol, HDL-C, LDL-C, triglyceride, very low-density lipoprotein, LDL, chylomicron), apolipoprotein AI, apolipoprotein AII,apolipoprotein B48, apolipoprotein CIII and apolipoprotein E, free fatty acids 1.4 waist circumference, hip circumference, waist/hip ratio

Safety

1. Safety of the study by comparing with conventional therapy, monitoring blood pressure, pulse rate, hematological parameters and urinalysis

DETAILED DESCRIPTION:
Subjects and methods Study product The test product is the pure D-allulose which is a rare sugar. The control product is the non-calorie sweetener erythritol.

Study design This is a single center, prospective, randomized, control trial. After informed consent is obtained, history taking and physical examination will be performed to ensure that the patients met all inclusion criteria and had no exclusion criteria.

At the screening day, venous blood samples will be collected following an overnight fasting of at least 8 hours. Complete blood count (CBC), chemistry including fasting plasma glucose (FPG), glycated hemoglobin (HbA1c), insulin, blood urea nitrogen (BUN), creatinine, lipid profiles (total cholesterol, HDL-C, LDL-C, triglyceride, very low-density lipoprotein), blood urea nitrogen, creatinine, total protein, Albumin, albumin/globulin ratio, glutamine oxaloacetic transaminase (GOT), glutamic pyruvic transaminase (GPT) , Gamma-glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), total bilirubin (including Direct and Indirect), alkaline phosphatase, uric acid, plasma amylase, cholinesterase, Sodium, Chloride, potassium, carbon dioxide , Calcium, inorganic phosphate, magnesium, plasma iron will be measured.

Urine will be collected for urinalysis and urine pregnancy test will be performed to exclude pregnant women from the study.

Visceral fat area (VFA), subcutaneous fat area (SFA), total fat area (TFA) will be measured with abdominal CT scan at umbilical level (L4) and bioelectrical impedance at D-7 or screening visit.

The eligible subjects will be randomized with an equal probability of receiving either pure D-allulose 5 g 3 times a day from 30 min before meal to right after meals (with any liquid) plus conventional therapy or placebo (non-calorie sweetener erythritol) 5 g 3 times a day from 30 min before meal to right after meal (with any liquid) plus conventional therapy for 24 weeks. Both the subjects and the investigator will be blinded to the type of the product. Subjects in both groups will be instructed to modify their lifestyle to control their diet to 1200 kcal for women and 1500 kcal for men and increase physical activity.

Subjects will be asked to do 3-d food record per week (2 working days and 1 weekend) entire of the study. Subjects will need to record any exercise they do including type and duration during in the study. Subjects will be asked to visit every 4 weeks for follow-up for totally 9 visits including screening day or D -7, D0, end of week 4, 8, 12, 16, 20, 24 and 4 weeks post intervention (at the end of week 28) in 29 weeks duration.

Assessment of insulin resistance index (IRI) was calculated from the homeostasis model assessment of insulin resistance (HOMA-IR) using FPG (mmol/L) multiply by fasting insulin (U/ml) divided with 22.5.

The satisfaction of the product will be asked at 4 weeks, 12 weeks and 24 weeks after consumption of the study products.

From the visit 1 to visit 8, same blood samples as the screening will be measured.

At the screening visit, visit 4 and visit 7, CT abdomen measurements will be conducted.

At the visit 1 and visit 7, adiponectin, leptin, tumor necrosis factor -alpha will be measured.

At the visit 1, visit 4, visit 7 and visit 8, other lipid profiles will be measured including very low-density lipoprotein and Chylomicron fractionation , Apolipoprotein (AI, AII，C-III, E), Apolipoprotein (B48, B100), nonesterified fatty acid

Adverse Event Assessment At each visit, subjects will be asked an open question as if he/she has experienced any abnormal symptoms. Any symptom reported by the subject will be recorded as an adverse events with details of the event, its severity, start and stop dates, and relationship to study products.

Withdrawal criteria

1. Consume study product less than 90% during treatment period
2. Start taking any medication that may affect body weight during in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years and legal age of consent.
2. If female, the subject is either post-menopausal or surgically sterilized, or has a negative urine pregnancy test within 7 days prior to enrollment and will use adequate contraception during the study.
3. Obesity, defined as BMI ≥ 25 kg/m2
4. Stable weight (weight change no more than 5% within 3 months)
5. If subject has been treated with medications that might cause weight change (such as corticosteroid, antidepressant, antipsychotics, oral contraceptive pills) prior to admission, he/she must have taken the medication regularly at a steady dose for at least 8 weeks up.
6. The subject has provided written informed consent prior to admission to the study.

Exclusion Criteria:

A subject will be excluded from the study for any of the following reasons:

1. Pregnancy or lactation
2. Diagnosed with diabetes mellitus
3. Weight change ≥ 5 % within 3 months prior to admission to the study
4. Has taken any weight loss medications within 3 months prior to admission to the study
5. Immunocompromised status, including a debilitated state or malignancy
6. Active liver, renal, thyroid diseases
7. Frequent alcoholic consumption more than twice a week; with beer > 360 mL, alcohol > 45 mL, wine > 150 mL for female, or beer > 720 mL, whisky > 90 mL, wine > 300 mL for male each time
8. Has gastrointestinal symptoms such as nausea, vomiting, loss of appetite, premature satiety, diarrhea, or chronic constipation
9. Lack of ability or willingness to give informed consent
10. Taken any medications than might cause weight loss or weight gain such as corticosteroid, antidepressant, antipsychotics, oral contraceptive pills < 8 weeks or change the dose of these medication with 8 week prior to admission
11. Enrolled in any other clinical study within 3 months before enrolment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Body composition change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Body weight change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
BMI change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Body fat percentage change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)

SECONDARY OUTCOMES:
insulin resistance change (as calculated from HOMA-IR) after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Fasting plasma glucose change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
HbA1c change after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Change in inflammatory markers (adiponectin, leptin and tumor necrosis factor-alpha) after 24 weeks of D-allulose consumption to erythritol consumption | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Change in lipid profiles | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Changes on waist circumference, hip circumference | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Changes on waist/ hip ratio | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)
Adverse events by monitoring clinical and laboratory data | 28 weeks (assess 4 weeks after 24 weeks consumption of the study product)

CONTACTS AND LOCATIONS:
Overall Officials: Supawan Buranapin, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Faculty of Medicine, Chiang Mai University, Muang Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cree GM, Perlin AS. O-isopropylidene derivatives of D-allulose (D-psicose) and D-erythro-hexopyranos-2,3-diulose. Can J Biochem. 1968 Aug;46(8):765-70. doi: 10.1139/o68-117. No abstract available. PMID 4299740
- [Background] Takeshita K, Suga A, Takada G, Izumori K. Mass production of D-psicose from d-fructose by a continuous bioreactor system using immobilized D-tagatose 3-epimerase. J Biosci Bioeng. 2000;90(4):453-5. doi: 10.1016/s1389-1723(01)80018-9. PMID 16232889
- [Background] Granstrom TB, Takata G, Tokuda M, Izumori K. Izumoring: a novel and complete strategy for bioproduction of rare sugars. J Biosci Bioeng. 2004;97(2):89-94. doi: 10.1016/S1389-1723(04)70173-5. PMID 16233597
- [Background] Matsuo T, Suzuki H, Hashiguchi M, Izumori K. D-psicose is a rare sugar that provides no energy to growing rats. J Nutr Sci Vitaminol (Tokyo). 2002 Feb;48(1):77-80. doi: 10.3177/jnsv.48.77. PMID 12026195
- [Background] Matsuo T, Izumori K. d-Psicose Inhibits Intestinal alpha-Glucosidase and Suppresses the Glycemic Response after Ingestion of Carbohydrates in Rats. J Clin Biochem Nutr. 2009 Sep;45(2):202-6. doi: 10.3164/jcbn.09-36. Epub 2009 Aug 28. PMID 19794929 (Retraction: PMID 24895485 J Clin Biochem Nutr. 2014 May;54(3):219)
- [Background] Iida T, Kishimoto Y, Yoshikawa Y, Hayashi N, Okuma K, Tohi M, Yagi K, Matsuo T, Izumori K. Acute D-psicose administration decreases the glycemic responses to an oral maltodextrin tolerance test in normal adults. J Nutr Sci Vitaminol (Tokyo). 2008 Dec;54(6):511-4. doi: 10.3177/jnsv.54.511. PMID 19155592
- [Background] Hayashi N, Iida T, Yamada T, Okuma K, Takehara I, Yamamoto T, Yamada K, Tokuda M. Study on the postprandial blood glucose suppression effect of D-psicose in borderline diabetes and the safety of long-term ingestion by normal human subjects. Biosci Biotechnol Biochem. 2010;74(3):510-9. doi: 10.1271/bbb.90707. Epub 2010 Mar 7. PMID 20208358
- [Background] Hossain A, Yamaguchi F, Matsunaga T, Hirata Y, Kamitori K, Dong Y, Sui L, Tsukamoto I, Ueno M, Tokuda M. Rare sugar D-psicose protects pancreas beta-islets and thus improves insulin resistance in OLETF rats. Biochem Biophys Res Commun. 2012 Sep 7;425(4):717-23. doi: 10.1016/j.bbrc.2012.07.135. Epub 2012 Aug 1. PMID 22877751
- [Background] Ochiai M, Onishi K, Yamada T, Iida T, Matsuo T. D-psicose increases energy expenditure and decreases body fat accumulation in rats fed a high-sucrose diet. Int J Food Sci Nutr. 2014 Mar;65(2):245-50. doi: 10.3109/09637486.2013.845653. Epub 2013 Oct 21. PMID 24144428
- [Background] Matsuo T, Izumori K. Effects of dietary D-psicose on diurnal variation in plasma glucose and insulin concentrations of rats. Biosci Biotechnol Biochem. 2006 Sep;70(9):2081-5. doi: 10.1271/bbb.60036. Epub 2006 Sep 7. PMID 16960391
- [Background] Ochiai M, Nakanishi Y, Yamada T, Iida T, Matsuo T. Inhibition by dietary D-psicose of body fat accumulation in adult rats fed a high-sucrose diet. Biosci Biotechnol Biochem. 2013;77(5):1123-6. doi: 10.1271/bbb.130019. Epub 2013 May 7. PMID 23649241
- [Background] Chung YM, Hyun Lee J, Youl Kim D, Hwang SH, Hong YH, Kim SB, Jin Lee S, Hye Park C. Dietary D-psicose reduced visceral fat mass in high-fat diet-induced obese rats. J Food Sci. 2012 Feb;77(2):H53-8. doi: 10.1111/j.1750-3841.2011.02571.x. PMID 22339545
- [Background] Wong JM, de Souza R, Kendall CW, Emam A, Jenkins DJ. Colonic health: fermentation and short chain fatty acids. J Clin Gastroenterol. 2006 Mar;40(3):235-43. doi: 10.1097/00004836-200603000-00015. PMID 16633129
- [Background] Haslam DW, James WP. Obesity. Lancet. 2005 Oct 1;366(9492):1197-209. doi: 10.1016/S0140-6736(05)67483-1. PMID 16198769
- [Background] The Western Pacific Region, World Health Organization, International Associates for the study of obesity, International Obesity Task Force. The Asia-Pacific Perspective: redefining obesity and its treatment. Melbourne: Health Communications Australia, 2000.
- [Background] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Background] Johnson WD, Brashear MM, Gupta AK, Rood JC, Ryan DH. Incremental weight loss improves cardiometabolic risk in extremely obese adults. Am J Med. 2011 Oct;124(10):931-8. doi: 10.1016/j.amjmed.2011.04.033. PMID 21962313